CLINICAL TRIAL: NCT00303589
Title: A Phase II Prospective, Open Label, Randomized, Active-controlled, Parallel Group, Multi-center 'Proof of Concept' Trial in Adult Patients With Complicated Skin or Skin Structure Infections Requiring Hospitalization.
Brief Title: A Study of Beta-Lactam in Hospitalized Patients With Skin and Skin Structure Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WI18274
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Soft Tissue Infections
MeSH Terms: conditions — Soft Tissue Infections | interventions — Standard of Care; beta-Lactams

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: beta-lactam
- 2 (Experimental)
  Interventions: Drug: beta-lactam
- 3 (Active Comparator)
  Interventions: Drug: Standard care

INTERVENTIONS:
Drug: Standard care — As prescribed
  Arms: 3
Drug: beta-lactam — 750mg iv q8h
  Arms: 1
Drug: beta-lactam — 1500mg iv q8h
  Arms: 2

SUMMARY:
This 3 arm study will compare the efficacy and safety of beta-lactam with that of 'standard care' in patients with complicated skin and skin structure infections requiring hospitalization. Patients will be randomized to receive 1)beta-lactam 750mg iv q8h 2)beta-lactam 1500mg iv q8h or 3)'standard care' [PRP (nafcillin or flucloxacillin) or vancomycin, plus aztreonam or ciprofloxacin]. The anticipated time on study treatment is <3 months and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* skin or skin structure infection requiring hospitalization;
* clinical diagnosis of a skin or skin structure infection caused by bacteria known or suspected to be susceptible to the randomized study treatment;
* material from site of infection is clinically purulent or seropurulent.

Exclusion Criteria:

* presenting with sustained shock (SBP<90mm Hg for > 2 hours, despite adequate fluid resuscitation);
* known or suspected concomitant bacterial infection requiring antibiotic treatment;
* skin infection or chronic non-healing ulcer of > 2 weeks duration;
* patients in whom surgery is the primary treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2005-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Clinical cure rate. | Event driven

SECONDARY OUTCOMES:
Time to clinical cure | Event driven
Time to resolution of signs and symptoms of skin or soft tissue infection | Event driven
Bacteriological outcome | Event driven
Adverse events; laboratory abnormalities | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (47):
- United States (7):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Melbourne, Florida
  - Miami Beach, Florida
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Winston-Salem, North Carolina
- Argentina (10):
  - Buenos Aires
  - Ciudadela
  - Córdoba
  - El Palomar
  - Entre Ríos
  - Granadero Baigorria
  - Merlo
  - Neuquén
  - Rosario
  - Santa Fe
- Bulgaria (4):
  - Pleven
  - Plovdiv
  - Sofia
  - Varna
- Estonia (2):
  - Tallinn
  - Tartu
- Germany (4):
  - Lübeck
  - Mainz
  - München
  - Münster
- Hungary (2):
  - Budapest
  - Győr
- Latvia (2):
  - Liepāja
  - Riga
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Peru (2):
  - La Victoria, Lima
  - Lima
- Romania (4):
  - Bucharest
  - Cluj-Napoca
  - Constanța
  - Târgu Mureş
- South Africa (7):
  - Benoni
  - Cape Town
  - Middleburg
  - Port Elizabeth
  - Pretoria
  - Sommerset West
  - Themba